CLINICAL TRIAL: NCT02295683
Title: Renal Sympathetic Denervation by Iberis System in Patients With Uncontrolled Hypertension - IBERIS - HTN Registry
Brief Title: Renal Sympathetic Denervation by Iberis System in Patients With Uncontrolled Hypertension - Iberis-HTN Registry
Acronym: Iberis
Status: Terminated | Type: Observational
Why Stopped: The study was prematurely discontinued due to the low rate of enrollment.
Sponsor: Terumo Europe N.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: T124E2
Record Dates: First submitted 2014-11-17; First posted 2014-11-20 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Resistant Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Renal Denervation

SUMMARY:
The purpose of this study is to document safety and efficacy of renal sympathetic denervation treatment in subjects with uncontrolled hypertension by using Iberis renal denervation system.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, single-arm, non-interventional and open-label registry to collect descriptive data from patients who receive renal sympathetic denervation treatment in accordance with routine hospital practice using Iberis system.

This registry will collect data prospectively from patients that receive renal sympathetic denervation treatment with use of Iberis renal denervation system and treatment will be applied according to the routine hospital practice. No additional tests are required specific to this registry. The registry will serve as a tool to collect clinical data in order to expand the knowledge base of safety, efficacy and functionality of the Iberis system in patients with resistant hypertension.

A minimum of 30 patients will be enrolled in Europe

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years or minimum age as required by local regulations.
* Patient has been thoroughly informed about this registry and signed Informed Consent Form.
* Patient with true resistant hypertension defined as:

  * Office systolic BP higher than 160 or 150mmHg in case of type 2 diabetes
  * Ambulatory BP with average BP>130mmHg or mean daytime>135mmHg in more than 70% of the measurements.
* Patients should be on stable hypertension therapy for at least 8 weeks before procedure, including spironolactone if they are supposed to be respondent as indicated by the specialized center/excellence unit on hypertension.

Exclusion Criteria:

* Previous renal artery intervention (balloon angioplasty or stenting).
* Evidence of renal artery atherosclerosis (defined as a renal artery stenosis >50%).
* Main renal arteries of less than 4mm diameter or less than 20mm in length.
* Presence of multiple main renal arteries in either kidney.
* Estimated glomerular filtration rate <45ml/min per 1,73m2
* Recent myocardial infarction, unstable angina pectoris or cerebrovascular accident within the past 3-6 months.
* False resistant hypertension (pseudo resistance) by using 24h ambulatory BP monitoring (ABPM).
* Secondary arterial hypertension.
* Pregnancy.
* There is another pathological process with well-known life expectancy of less than 5 years.
* Patient unable to do correct FU.
* Unable to take correct ambulatory BP.
* Primary hyperaldosteronism.
* Known lack of adherence to medical treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with uncontrolled hypertension entitled to receive renal sympathetic denervation treatment per routine hospital practice and according to relevant international, or country specific guidelines
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2014-11; Primary Completion 2016-11-30 (Actual); Study Completion 2017-09-04 (Actual)

PRIMARY OUTCOMES:
Blood Pressure (BP) Measurements | Up to 5 year FU
  Office BP; Ambulatory BP; Home BP

CONTACTS AND LOCATIONS:
Overall Officials: José Ramon Rumoroso, Dr., Principal Investigator — Hospital Galdakao; Palop López, Dr., Principal Investigator — Hospital San Juan Alicante; Mauri, Dr., Principal Investigator — Germans Trias i Pujol Hospital; Perez, Dr., Principal Investigator — Hospital de Léon; Garcia, Dr., Principal Investigator — Hospital Monteprincipe; Goicolea, Dr., Principal Investigator — Hospital Puerta de Hierro; Goran Stankovic, Dr., Principal Investigator — Clinical Center of Serbia
Locations (2):
- Clinical Center of Serbia, Belgrade, Serbia
- Hospital Galdakao, Galdakao, Spain